CLINICAL TRIAL: NCT07232862
Title: Analysis Of The Effect Of A Fine Manual Skills Intervention In A Specific Context On The Linguistic Processing of Healthy Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mandala
Record Dates: First submitted 2025-09-12; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Context-Specific Fine Motor Skills Training (Experimental)
  Interventions: Behavioral: Context-Specific Fine Motor Skills Training
- Fine Motor Skills Training (Active Comparator)
  Interventions: Behavioral: Fine Motor Skills Training

INTERVENTIONS:
Behavioral: Context-Specific Fine Motor Skills Training — The intervention for the "Context-Specific Fine Motor Skills Training" group will consist of practicing fine manual dexterity in a task-oriented context, characterized by clear and functional objectives. The activity will begin with solving mathematical calculations, the results of which will range from 1 to 4, each associated with a specific color of bead. Using tweezers, the participant must select the bead corresponding to the result obtained, apply glue, and fill the indicated space of the mandala. The intervention will be carried out for 20 minutes per day, five times a week, over the course of two weeks.
  Arms: Context-Specific Fine Motor Skills Training
Behavioral: Fine Motor Skills Training — The "Fine Motor Skills Training" group will undergo an intervention with a less complex task. Participants will complete the mandala using only their hands to manipulate the beads. The duration and frequency protocol will be identical to that of the experimental group, with 20-minute sessions, five times a week, over two weeks.
  Arms: Fine Motor Skills Training

SUMMARY:
This is a randomized, single-blind clinical trial that will include healthy individuals between the ages of 19 and 24. Participants with previously diagnosed neurological and/or psychiatric disorders, a history of traumatic brain injury, use of psychoactive substances or medications that may affect cognition, and pregnant women or women suspected of being pregnant will be excluded. The sample will be a convenience sample, with participants randomly allocated to intervention and control groups (1:1), and the sample size calculation will be based on a pilot study. Participants will be assessed at two different time points, before and after the intervention, for fine manual dexterity and syntactic language processing. The intervention group will undergo fine manual dexterity training in a specific context, while the control group will undergo an intervention with a less complex task and without a specific context. Both protocols will consist of 20-minute sessions, held five times a week over two weeks, in a synchronous online format, via the Google Meet videoconferencing platform.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed young people between 19 and 24 years old;
* Accept participation in the study and sign the free and informed consent form.

Exclusion Criteria:

* Presence of previously diagnosed neurological and/or psychiatric disorders;
* History of traumatic brain injuries;
* Pregnant women or women suspected of being pregnant.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-13 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive effort | Baseline (2 to 3 days before the beginning of intervention) and post-intervention (2 weeks after the beginning of intervention, and 1 day after the last day of intervention)
  Cognitive effort will be assessed through EEG by analyzing activity in the Theta, Alpha, and Beta frequency bands. Increases in frontal Theta indicate higher cognitive demand, reductions in parietal Alpha reflect greater attentional engagement, and increases in Beta are associated with heightened mental activation during complex tasks. These patterns allow for an objective identification of the cognitive load involved.

SECONDARY OUTCOMES:
Syntactic processing | Baseline (2 to 3 days before the beginning of intervention) and post-intervention (2 weeks after the beginning of intervention, and 1 day after the last day of intervention)
  Our research team developed a Syntactic Processing Assessment consisting of 180 sentences, divided into three categories: 60 sentences with gender violation, 60 sentences with number violation, and 60 "control" sentences that do not have any syntactic error. That test will be administered through a program developed in the Python language, where the participant will have 400ms to respond to each sentence: correct or incorrect.
Fine motor dexterity | Baseline (2 to 3 days before the beginning of intervention) and post-intervention (2 weeks after the beginning of intervention, and 1 day after the last day of intervention)
  The fine motor dexterity will be evaluated through the Grooved Pegboard Test. The test consists of picking a pine and putting it in the pegboard in a correct sequence. The pegboard had 25 holes, and the score is measured in how much time the participant spends completing the pegboard.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UFCSPA, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided